CLINICAL TRIAL: NCT05432609
Title: Standardization and Reproducibility Regarding Scanning Procedures and Measurements of Weight-bearing Cone Beam CT in the Lower Extremity
Status: Active, not recruiting | Type: Observational
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Signe Brinch, Principal investigator, MD, PhD student, Bispebjerg Hospital
Other Study IDs: H-20068116
Record Dates: First submitted 2022-06-21; First posted 2022-06-27 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Musculoskeletal Diseases
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Healthy: Weight bearing CT in fully extended and flexed (20 degrees) position, loaded and unloaded, respectively.
  Interventions: Diagnostic Test: Weight bearing CT
- Trochlear dysplasia: Weight bearing CT in fully extended and flexed (20 degrees) position, loaded and unloaded, respectively.
  Interventions: Diagnostic Test: Weight bearing CT

INTERVENTIONS:
Diagnostic Test: Weight bearing CT — Weight bearing CT in loaded and unloaded positions

SUMMARY:
Cone Beam CT (CBCT) of the knee is gaining interest, especially regarding patients suffering from patellofemoral instability. With this study investigators wish to investigate the day-to-day, test-retest reliability of weight bearing (WB) and non-weight bearing (NWB) CBCT of the knee in healthy participants and patients suffering from trochlear dysplasia. The participants and patients will be scanned in the following positions: 0° WB, 0° NWB, 20° WB, 20° NWB on two separate days. The trochlear dysplasia patients will furthermore be scanned 6 months postoperatively.

The aim is to develop af protocol on how to both position patients during weight bearing scannings as well as a protocol on how to prepare the cross sectional images before measurements.

DETAILED DESCRIPTION:
Investigators expect that scans performed with CBCT will show a clear change in the TT-TG distance when comparing scans performed in two different degrees of flexion of the knee. Investigators expect a discrete change in the TT-TG distance between non-weight bearing and weight-bearing state of the same degree of flexion. Investigators expect that other radiological targets for assessing patellofemoral instability, e.g. in trochlear dysplasia patients will change between the different scan situations. In addition, investigators expect that the TT-TG distance measurement method has a high reproducibility of intra- and in-terobserver variation as well as over time with repeated scans. The reproducibility is expected to be at least as good or above existing 2D measurement methods on conventional scans. In patients with trochlear dysplasia, a greater TT-TG distance is expected than in healthy controls. In addition, differences in TT-TG distance between flexion/extension as well as between non-weight bearing and weight bearing condition are expected to be greater than in healthy controls. In addi-tion, investigators expect to be able to detect a correlation between controlled changes in the position of the foot which will lead to passive changes in the TT-TG distance.

The purpose of the study is:

* To investigate changes in TT-TG distance in CBCT scans of the knee joint, in healthy con-trols as well as in trochlear dysplasia patients, in two predefined degrees of flexion (0 ° i.e. fully stretched position; 20 ° flexion), in respectively weight-bearing loaded and unloaded position
* To investigate the day-to-day reliability of the measured TT-TG distance, knee flexion angle and other radiological measurements regarding patellofemoral instability, at two separate CBCT scan sessions in patients with trochlear dysplasia compared with healthy controls
* To investigate changes in the TT-TG distance in trochlear dysplasia patients before and after surgery in terms of evaluation of the patellofemoral instability

ELIGIBILITY:
Inclusion Criteria:

Substudy 1:Healthy

* Male or female aged 18-39 years
* Must be able to stand on one leg for 30 seconds

Substudy 2

* Diagnosed with trochlear dysplasia, in addition healthy
* Male or female aged 18-39 years
* Patients scheduled to either a trochlear plastic surgery + MPFL reconstruction or Elmslie- Trillat + MPFL reconstruction + trochlear plastic surgery
* Must be able to stand on one leg for 30 seconds

Exclusion Criteria:

Substudy 1

* Current knee injury and / or knee pain.
* Known rheumatoid and / or connective tissue disease.
* Previous treatment requiring knee injury and / or knee surgery.
* Pregnancy

Substudy 2

* Known rheumatoid and / or connective tissue disease
* Previous treatment requiring knee injury and / or knee surgery.
* Patients who need distalization
* Pregnancy

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy participants recruited amongst employees in the ER, Bispebjerg-Frederiksberg Hospital Trochlear dysplasia patients selected from the sports surgery unit, Bispebjerg-Frederiksberg Hospital
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
Measurement of patellofemoral indices | 1 year
  Intra and interrater reliability and day to day repeatability

CONTACTS AND LOCATIONS:
Overall Officials: Signe Brinch, MD, Principal Investigator — University Hospital Bispebjerg and Frederiksberg
Locations (1):
- Dept. of Radiology, Bispebjerg-Frederiksberg Hospital, Copenhagen, Denmark